CLINICAL TRIAL: NCT05722418
Title: A Phase 1, Multicenter, Open-Label Study of CB-011, a CRISPR-Edited Allogeneic Anti-BCMA CAR-T Cell Therapy in Patients With Relapsed/Refractory Multiple Myeloma (CaMMouflage Trial)
Brief Title: CRISPR-Edited Allogeneic Anti-BCMA CAR-T Cell Therapy in Patients With Relapsed/Refractory Multiple Myeloma
Acronym: CaMMouflage
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Caribou Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CB11A
Record Dates: First submitted 2022-12-19; First posted 2023-02-10 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-08

CONDITIONS: Relapsed/Refractory Multiple Myeloma
Keywords: CaMMouflage; Allogeneic; Multiple Myeloma; Relapse Refractory Multiple Myeloma; CAR-T Cells; BCMA; Cell Therapy; Cellular Immuno-therapy; CB11A; CB-011; CB-011A; CAR-T; Anti BCMA; ALLO CAR T
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CB-011 (Experimental): * Part A Escalation with CB-011 in ascending doses using a traditional 3+3 design.
  * Part B Expansion. Up to 30 participants will be enrolled to receive CB-011 at the RDE/MTD and/or RP2D determined in Plan A
  Interventions: Biological: CB-011

INTERVENTIONS:
Biological: CB-011 — CB-011 allogeneic CAR T cell therapy targeting BCMA Cyclophosphamide Chemotherapy for lymphodepletion Fludarabine Chemotherapy for lymphodepletion
  Other Names: Cyclophosphamide; Fludarabine

SUMMARY:
This is a Phase 1 study to evaluate the safety of CB-011 (the study treatment), an allogeneic chimeric antigen receptor (CAR-T) cell therapy that targets the B cell maturation antigen (BCMA), to determine the best dose of CB-011, and to assess the effectiveness of CB-011 in treating multiple myeloma that has come back (relapsed) or that is no longer responding to other treatment (refractory).

ELIGIBILITY:
Inclusion Criteria:

1. Documented diagnosis of relapsed/refractory multiple myeloma (MM) with measurable disease (according to IMWG diagnostic criteria.)
2. Received at least 3 prior MM treatment lines of therapy which must include a proteasome inhibitor (PI), an immunomodulatory drug (IMiD), and an anti-CD38 monoclonal antibody as part of a prior line of therapy, either in monotherapy or in combination.
3. Eastern Cooperative Oncology Group performance status grade of 0 or 1.
4. Adequate hematologic, renal, hepatic, pulmonary, and cardiac function.

Exclusion Criteria:

1. Prior treatment with CAR-T cell therapy directed at any target.
2. Autologous stem cell transplant within the last 6 weeks before lymphodepletion.
3. Allogeneic stem cell transplant within 6 months before lymphodepletion.
4. Known active or prior history of CNS involvement.
5. Stroke or seizure within 6 months of signing ICF.
6. Seropositive for or history of human immunodeficiency virus.
7. Vaccinated with live, attenuated vaccine within 4 weeks prior to lymphodepletion.
8. Hepatitis B infection.
9. Hepatitis C infection.
10. Known life-threatening allergies, hypersensitivity, or intolerance to CB-011 or its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
(Part A) Number of patients with dose limiting toxicities (DLT) | 28 days
  Number of patients with DLTs during the 28 days following the first administration of CB-011.
(Part B) Overall Response Rate (ORR) | 12 Months
  The ORR will be evaluated by International Myeloma Working Group (IMWG) criteria.

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - CU Anschutz Medical Campus, Anshutz Cancer Pavillion, Aurora, Colorado
  - Sylvester Comprehensive Cancer Center, University of Miami Hospital and Clinics, Miami, Florida
  - University of Kentucky/ Markey Cancer Center, Lexington, Kentucky
  - Hackensack Meridian John Theurer Cancer Center, Hackensack, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Health System (DUHS), Durham, North Carolina
  - Oncology Hematology Care, Inc, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Tennessee Oncology, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin